CLINICAL TRIAL: NCT01599572
Title: Zinc Intervention in Nursing Home Elderly
Brief Title: Effect of Zinc Supplementation on Serum Zinc Level in Nursing Home Elderly
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: Boston University (Other); Hebrew SeniorLife (Other); Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 8541
Record Dates: First submitted 2012-05-14; First posted 2012-05-16 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Disorder of Immune Function
Keywords: zinc supplementation; serum zinc concentration; lymphocyte proliferation
MeSH Terms: conditions — Immune System Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- 30mg/day zinc supplementation (Experimental): 30mg/day of zinc supplement provided for 3 months to zinc deficient elderly
  Interventions: Other: zinc supplementation

INTERVENTIONS:
Other: zinc supplementation — 30mg/day of zinc in the form of zinc gluconate
  Other Names: zinc was provided in the form of zinc gluconate

SUMMARY:
Background: Zinc supplementation has the potential to improve serum zinc levels and immunity of zinc deficient nursing home elderly.

Objective: To determine the effect of zinc supplementation of 30mg/d for 3 months on serum zinc levels and T-cell mediated function of zinc deficient nursing home elderly.

Design: This is a randomized, double-blind, placebo-controlled study. Outcome measures included change in serum zinc levels and various T-cell mediated immune factors between baseline and month 3.

Hypotheses: The investigators hypothesize that zinc supplementation of 30mg/d for 3 months will improve serum zinc levels as well as various T-cell mediated immune factors in zinc deficient nursing home elderly.

DETAILED DESCRIPTION:
Four hundred and forty-two medical charts were screened from three participating nursing homes; 53 nursing home elderly were eligible and therefore were screened for low serum zinc levels (<70µg/dL). Of these, 31 (58%) had low serum zinc levels. Participants were randomized into either the placebo (N=16) or the zinc supplemented (N=15) group. Six participants did not complete the study for various reasons including refusal to take study capsules, and advice from their physicians; one participant in the zinc group experienced nausea on two consecutive days following ingestion of the zinc capsule at the beginning of the study. A total of 25 participants completed the study with 13 and 12 receiving the placebo and zinc capsules, respectively, over a period of three months

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥65 years of age.
2. More than 6 months life expectancy, in the judgment of their study physician.
3. Willing to be randomized to one of the treatment groups.
4. Able to swallow pills.
5. Not currently on antibiotics.
6. Subjects consuming DRI levels of supplements and willing to replace their supplement with our control supplement.
7. Supplements of calcium, vitamin D, and iron will be permitted.
8. Willing to receive influenza vaccine.

Exclusion Criteria:

1. Anticipated transfer or discharge within three months of enrollment.
2. Bed- or room-bound continuously for the last three months.
3. Presence of lung neoplastic diseases or other active neoplastic diseases requiring chemotherapy and/or use of immunosuppressive drugs (including no more than 10 mg/day of prednisone).
4. Naso-gastric or other tube feeding.
5. Long-term intravenous or urethral catheters (30 days).
6. Presence of tracheostomy or chronically ventilator-dependent.
7. Consuming supplements containing more than the DRI level of nutrients known to affect the immune response, i.e. vitamins E, C, B6, selenium, zinc, or β -carotene and unwilling to stop.
8. Chronic prophylactic antibiotic treatment (low percent of subjects meeting other inclusion criteria). 9) Protein energy malnutrition defined as albumin < 3.0 g/dl and BMI <18 kg/m2.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-07; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
serum zinc concentration | 3 months

SECONDARY OUTCOMES:
lymphocyte proliferation | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Simin N Meydani, DVM, PhD, Principal Investigator — HNRCA-tufts University